CLINICAL TRIAL: NCT05192135
Title: Influence of Hematocrit Level on the Visibility of the Venous Network in Magnetic Susceptibility Imaging
Acronym: HEMAT_SWI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: HEMAT_SWI
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Magnetic susceptibility imaging is a magnetic resonance imaging (MRI) technique that uses the magnetic properties of tissues and the BOLD (blood oxygen level-dependent) effect. It allows a better visualization of venous structures and hemorrhagic lesions. These sequences are now used in clinical routine.

The extreme sensitivity of these sequences to the oxy/deoxyhemoglobin ratio makes it possible to describe a new MRI semiology, particularly in the context of cerebral ischemia. The interest of the analysis of the venous network signal, which can reflect cerebral perfusion, has been reported.

However, the influence of the hematocrit level on the signal of the venous network in magnetic susceptibility imaging has not been evaluated at present. It seems important to better define the influence of hematocrit level on the signal of the veins with this sequence to avoid potential diagnostic errors.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient referred to GHPSJ for suspected stroke
* Patient who had a brain MRI including the magnetic susceptibility sequence
* Patient for whom a blood count with hematocrit was performed at the same time (within 7 days between the MRI and the blood test)
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Elimination of potential biases: recent injection (48 h) of gadolinium, pathology likely to modify the venous signal in magnetic susceptibility imaging (notably arterial occlusion or stenosis), high flow oxygenation, sickle cell disease, thalassemia.
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients were referred for suspected stroke, between January 1, 2016, and May 1, 2021. who had a brain MRI including the magnetic susceptibility sequence Patients for whom a blood count with hematocrit was performed at the same time (within a 7-day interval between the MRI and the blood test).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific influence of the hematocrit level on the visibility of the venous network | Day 1
  This outcome corresponds to the visibility of the venous network in magnetic susceptibility imaging using a visual scale allowing comparison between patients with normal hematocrit, anemia or polycythemia.

SECONDARY OUTCOMES:
Inter-observer agreement of the visual analysis of the venous network | Day 1
  This outcome corresponds to the correlation of visual scales between different observers.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah TOLEDANO, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Haacke EM, Mittal S, Wu Z, Neelavalli J, Cheng YC. Susceptibility-weighted imaging: technical aspects and clinical applications, part 1. AJNR Am J Neuroradiol. 2009 Jan;30(1):19-30. doi: 10.3174/ajnr.A1400. Epub 2008 Nov 27. PMID 19039041
- [Background] Mittal S, Wu Z, Neelavalli J, Haacke EM. Susceptibility-weighted imaging: technical aspects and clinical applications, part 2. AJNR Am J Neuroradiol. 2009 Feb;30(2):232-52. doi: 10.3174/ajnr.A1461. Epub 2009 Jan 8. PMID 19131406
- [Background] Chalian M, Tekes A, Meoded A, Poretti A, Huisman TA. Susceptibility-weighted imaging (SWI): a potential non-invasive imaging tool for characterizing ischemic brain injury? J Neuroradiol. 2011 Jul;38(3):187-90. doi: 10.1016/j.neurad.2010.12.006. Epub 2011 Feb 26. PMID 21354625
- [Background] Wang Y, Shi T, Chen B, Lin G, Xu Y, Geng Y. Prominent Hypointense Vessel Sign on Susceptibility-Weighted Imaging Is Associated with Clinical Outcome in Acute Ischaemic Stroke. Eur Neurol. 2018;79(5-6):231-239. doi: 10.1159/000488587. Epub 2018 Apr 19. PMID 29672289
- [Background] Horie N, Morikawa M, Nozaki A, Hayashi K, Suyama K, Nagata I. "Brush Sign" on susceptibility-weighted MR imaging indicates the severity of moyamoya disease. AJNR Am J Neuroradiol. 2011 Oct;32(9):1697-702. doi: 10.3174/ajnr.A2568. Epub 2011 Jul 28. PMID 21799039
- [Background] Winchell AM, Taylor BA, Song R, Loeffler RB, Grundlehner P, Hankins JS, Wang WC, Ogg RJ, Hillenbrand CM, Helton KJ. Evaluation of SWI in children with sickle cell disease. AJNR Am J Neuroradiol. 2014 May;35(5):1016-21. doi: 10.3174/ajnr.A3794. Epub 2013 Nov 21. PMID 24263696